CLINICAL TRIAL: NCT03944720
Title: Prospective Evaluation on the Efficacy of Transvaginal Repair for Rectocel
Brief Title: Efficacy of Transvaginal Repair for Rectocele
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment in participating centers
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: Hospital Universitari MútuaTerrassa (Unknown); Heling HartZiekenhuis Lier (Other); Hospital Clinico Universitario San Cecilio (Other)
Responsible Party: Principal Investigator, Yolanda Ribas, Principal investigator, Consorci Sanitari de Terrassa
Other Study IDs: 02-18-102-024
Record Dates: First submitted 2019-05-03; First posted 2019-05-09 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Rectocele; Surgery
MeSH Terms: conditions — Rectocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with rectoceles may present a variety of symptoms such as pelvic pressure, obstructive defecation or discomfort during sexual intercourse. The main symptom of the patient probably ends up conditioning if the patient is referred to a gynaecologist or a colorectal surgeon.

Different surgical techniques have been described to repair the rectocele. The posterior colporrhaphy is the preferred approach for most gynaecologists, while the transanal repair is the most common approach for the majority of colorectal surgeons. However, the small number of prospective studies, the inconsistent inclusion criteria and the variability of the outcome measures make difficult to know what the ideal surgical approach for a rectocele repair would be. Gynaecologists usually do not assess defecatory function before a rectocele repair, and studies focused on obstructive defecation include patients with other co-existing pathologies (rectal prolapse, rectal intussusception, enterocele) that may influence the success of the repair. Moreover, functional disorders such as the paradoxical contraction of the external anal sphincter or the puborectalis muscle are not systematically reported. On the other hand, many surgeons have questioned the transvaginal approach because it has been reported that patients may present dyspareunia after the surgery, although it is not systematically evaluated.

The hypothesis of the investigators is that the transvaginal approach for rectocele repair is an effective treatment for symptoms of obstructive defecation and is not associated with sexual dysfunction when the plication of the puborectalis muscle is not performed.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Older than 18 year old
* Symptoms of obstructed defecation associated to a rectocele with an indication for surgery according to the following criteria:

  1. Symptoms of obstructed defecation according to Rome III criteria: straining, sensation of incomplete evacuation, sensation of anorectal obstruction/blockage, and/or manual manoeuvres to facilitate defecation at least in 25% of defecations for the last 3 months
  2. Incomplete emptying of the rectocele on a defecography
  3. Failure of conservative treatment including dietary advice and laxatives, with persisting symptoms of obstructive defecation
  4. Recto-rectal intussusception may coexist on defecography (grade I and II of Oxford Prolapse Grading System)
  5. Non-obstructive enterocele may coexist on defecography (type A enterocele: the small bowel descends to puboccoccygeal line (PCL) during straining and returns to PCL at the end of the straining attempt without compressing the rectal ampulla or compressing it from above with no obstruction)
  6. Absence of anal sphincter dyssynergia on anorectal manometry, or successful rehabilitation after biofeedback in the case of previous dyssynergia
* Ability to understand the surgical procedure and the questionnaires of the study
* Written informed consent

Exclusion Criteria:

* Anal sphincter dyssynergia
* Coexisting recto-anal intussusception on defecography or external rectal prolapse (grades III, IV and V Oxford Prolapse Grading System)
* Coexisting enterocele compressing/obstructing the rectum on defecography (type B enterocele: the enterocele descends beyond the PCL to the perineum through the rectovaginal space to compress the rectal ampulla at the end of the evacuation process; type C enterocele (obstructive): the enterocele descends beyond the PCL to the perineum through the rectovaginal space to compress the rectal ampulla at the beginning of the evacuation process)
* Slow transit constipation associated to obstructed defecation
* Severe psychiatric disorder
* Refusal to provide written informed consent

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females may present with anterior rectocele
Study Population: Patients with indication for rectocele surgical repair fulfilling the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of obstructive defecation measured by the Altomare obstructed defecation syndrome (ODS) score | Baseline, 6 months and 12 months after surgery
  Assessment of the efficacy of the transvaginal approach for rectocele repair to improve symptoms of obstructive defecation according to the Altomare ODS score. The Altomare ODS score is a validated questionnaire to assess the severity of the obstructed defecation syndrome, consisting of eight 3- o 4-point Likert-scaled symptom items. Each of the items has four or five possible answers with scores ranging from zero (symptom free) to three or four points (more severe symptom). The ODS score is the sum of all points, with a maximum possible of 31 points.
Change in symptoms of obstructive defecation measured by the KESS score | Baseline, 6 months and 12 months after surgery
  Assessment of the efficacy of the transvaginal approach for rectocele repair to improve symptoms of obstructive defecation according to the KESS score. The KESS (Knowles-Eccersley-Scott-Symptom) score is a validated questionnaire to assist in diagnosing constipation and in discriminating among pathophysiologic subgroups, consisting of eleven questions. Each question has four to five possible answers which are scored on an unweighted linear integer scale to produce a range between zero and three, or zero and four points. Lower scores represent symptom-free states and higher scores, increased symptom severity. The KESS score is the sum of all points, with a maximum possible of 39 points.

SECONDARY OUTCOMES:
Changes in sexual function | Baseline, 6 months and 12 months after surgery
  To assess changes in the Female Sexual Function Index (FSFI) questionnaire. The FSFI score is a validated 19-item questionnaire to measure the sexual functioning in women, including six domains: desire, subjective arousal, lubrication, orgasm, satisfaction and pain. Domain scoring is as follows: desire 2-10, arousal 0-20, lubrication 0-20, orgasm 0-15, satisfaction 2-15, pain 0-15. Lower scores represent worse sexual functioning.
Assessment of morbidity related to the surgical technique | Baseline, 6 months and 12 months after surgery
  Description of the morbidity that may be related to any surgical technique

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
All data will be included in the same database and analyzed together